CLINICAL TRIAL: NCT06107972
Title: Developing a Culturally Adapted Intervention for Latino Youth Transitioning to Adulthood
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: UTHealth Houston Seed Grant and Autism Speaks Fellowship (Unknown)
Responsible Party: Principal Investigator, Antonio Pagan, Postdoctoral Research Fellow, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0188
Record Dates: First submitted 2023-10-22; First posted 2023-10-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Launching! to Adulthood (¡Iniciando! la Adultez) program (Experimental)
  Interventions: Behavioral: Launching! to Adulthood (¡Iniciando! la Adultez) program

INTERVENTIONS:
Behavioral: Launching! to Adulthood (¡Iniciando! la Adultez) program — The program includes cognitive behavioral and acceptance and commitment therapy, with a focus on developing goals during the transition to adulthood through a values framework. After a combined (parents and young adults) 90-minute introductory group meeting in-person, parents and the transition-aged young adults with ASD attend 9 separate, 90-minute weekly group telehealth meetings. Additionally, young adults have weekly personal coaching meetings for 30-minutes to discuss progress toward goals and barriers encountered. Leaders teach transition-aged young adult's skills through various social activities, as well as other skills (e.g., emotion regulation, cognitive diffusion) to help overcome barriers towards their goals. The treatment targets three core factors (i.e., mental health conditions, social skills, and coping with and adapting to stress). Leaders teach parents new parenting skills, knowledge of ASD, and readiness to support their young adult's transition to independent life.

SUMMARY:
The purpose of this study is to evaluate the acceptability, feasibility (e.g., satisfaction, completion rate, barriers to recruitment, treatment fidelity) of the culturally refined Launching! to Adulthood (¡Iniciando! la Adultez) program, to test for a preliminary signal of effect between baseline and post-treatment for the Launching! to Adulthood (¡Iniciando! la Adultez) program and to identify preliminary neural mechanisms of action, including biomarkers of brain structure and connectivity, in terms of treatment response for 15 Latino young adults participating in the ¡Iniciando! therapy program.

DETAILED DESCRIPTION:
The Launching! to Adulthood (¡Iniciando! la Adultez) program uses a culturally sensitive therapy program that was translated into Spanish to help Latino young adults with Autism Spectrum Disorder (ASD) who are transitioning to adulthood (18-25 years old) and their parents. The program aims to make the transition to adulthood easier for young adults and their families, and it includes specific cultural values of Latino young adults and their family members. The ¡Iniciando! la adultez program helps autistic young adults manage mental health needs like depression and anxiety and also addresses several areas impacting transition, including mental health barriers, executive functioning, and motivation. The ¡Iniciando! program also helps parents manage their own needs and addresses several areas, including psychoeducation and mental health.

ELIGIBILITY:
Inclusion Criteria:

* confirmed case of ASD
* a score of >14 on the Social Communication Questionnaire-Lifetime (SCQ-L110) completed with the mother or father
* meet DSM-5 criteria for ASD based on a Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 ASD symptom checklist
* previous diagnosis of ASD from a licensed mental health or medical professional
* speak English
* have a parent willing to participate
* score >85 on verbal intelligence quotient (IQ) on the Kaufman Brief Intelligence Test (KBIT-2)

Exclusion Criteria:

* history of a psychotic disorder or current psychotic symptoms
* suicidal ideation with intent or plan
* current alcohol or other substance use disorder rated severe
* concurrent enrollment in another clinical trial for autism spectrum disorder
* expression of unwillingness to complete study procedures
* For fMRI, unable to undergo fMRI scanning due to metallic devices or objects (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips, or other implanted metal parts) or claustrophobic to the scanner.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in adaptive behavior as assessed by the Adaptive Behaviour Assessment System, Third Edition | baseline, mid-treatment (5 weeks after baseline) , post-treatment (12 weeks after baseline), 3 month follow up, 6 month follow up
  This is a 239 item questionnaire and each is scored from 0(is not able to do this behavior) to 3 [(always able to do this behavior)(or almost always)] a higher number indicating better outcome
Change in Quality of life as assessed by the Autism Spectrum Quality of Life (ASQoL) questionnaire | baseline, mid-treatment (5 weeks after baseline) , post-treatment (12 weeks after baseline), 3 month follow up, 6 month follow up
  This is a 9 item questionnaire. Questions 1-5 and 9 are each scored from 1(not at all) to 5(totally) a higher number indicating better outcome and questions 6-8 are reverse scored from 5(never) to 1(always) a higher score indicating worse outcome
Change in Anxiety as assessed by the Generalized Anxiety Disorder-7 (GAD7) | baseline, mid-treatment(5 weeks after baseline) , post-treatment (12 weeks after baseline), 3 month follow up, 6 month follow up
  This is a 7 item questionnaire and each is scored from 0(not at all) to 4(nearly every day) for a maximum score of 21 , higher score indicating more anxiety
Change in depression as assessed by the Patient Health Questionnaire (PHQ-9) | baseline, mid-treatment(5 weeks after baseline) , post-treatment (12 weeks after baseline), 3 month follow up, 6 month follow up
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a maximum score of 27, higher number indicating worse outcome

SECONDARY OUTCOMES:
Change in caregiver burden as assessed by the Rapid Screen for Caregiver Burden (CBI) | baseline, mid treatment (5 weeks after baseline) , post-treatment (12 weeks after baseline), 3 month follow up, 6 month follow up
  This is a 24 item questionnaire, each item is given a score between 0 (not at all descriptive) and 4 (very descriptive), where higher scores indicate greater caregiver burden
Change in efficacy of coping with life's challenges as assessed by the Coping Self-Efficacy Scale (CSES) | baseline, mid treatment (5 weeks after baseline) , post-treatment (12 weeks after baseline),3 month follow up, 6 month follow up
  This is a 26 item questionnaire and each is scored on a 11-point scale from 0(cannot do at all)-10 (certain can do) and higher number indicates better outcome
Change in stress as assessed by the Riverside Acculturation Stress Inventory (RASI) | baseline, mid treatment (5 weeks after baseline) , post-treatment (12 weeks after baseline), 3 month follow up, 6 month follow up
  This is a 15-item scale and each is scored on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree) higher number indicates worse outcome
Change in goal attainment Goal Attainment Scaling (GAS) | week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12
  This is scored on a 5-point scale, with the degree of attainment captured for each goal area: If the patient achieves the expected level, this is scored at 0. If they achieve a better than expected outcome this is scored at: +1 (somewhat better) +2 (much better) If they achieve a worse than expected outcome this is scored at: -1 (somewhat worse) or -2 (much worse) Goals may be weighted to take account of the relative importance of the goal to the individual, and/or the anticipated difficulty of achieving it.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pagan, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No